CLINICAL TRIAL: NCT03245125
Title: Impacts of High-intensity Interval Training on Long-term Survival of Heart Failure Patients
Brief Title: HIIT Improves Survival of Heart Failure Patients
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 201601068B0
Record Dates: First submitted 2017-08-08; First posted 2017-08-10 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Heart Failure; Cardiac Rehabilitation; Cardiac Remodeling, Ventricular
MeSH Terms: conditions — Heart Failure; Ventricular Remodeling | interventions — High-Intensity Interval Training

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HIIT subjects in HFrEF patients: heart failure patients with reduced ejection fraction (HFrEF) received at least 36 times of high-intensity interval training (HIIT)
  Interventions: Behavioral: High-intensity interval training
- MDP subjects in HFrEF patients: heart failure patients with reduced ejection fraction (HFrEF) received only multidisciplinary disease management program (MDP) and underwent less than 36 times of high-intensity interval training (HIIT) or no exercise training
  Interventions: Behavioral: High-intensity interval training
- HIIT subjects in HFpEF patients: heart failure patients with preserved ejection fraction (HFpEF) received at least 36 times of high-intensity interval training (HIIT)
  Interventions: Behavioral: High-intensity interval training
- MDP subjects in HFpEF patients: heart failure patients with preserved ejection fraction (HFpEF) received only multidisciplinary disease management program (MDP) and underwent less than 36 times of high-intensity interval training (HIIT) or no exercise training
  Interventions: Behavioral: High-intensity interval training

INTERVENTIONS:
Behavioral: High-intensity interval training — Patients warmed up for 3 min at 30% of peak oxygen consumption (VO2peak). Five 3-minute intervals at 80% of VO2peak and each interval was separated by 3-minute exercise at 40% of VO2peak. The exercise session was terminated by 3-minute cool-down at 30% of VO2peak. All subjects used a EKG and BP monitors as indicators of the assigned exercise intensity. Borg 6-to-20 scale was used to assess the rate of perceived exertion during and after each exercise session. Patients suffering unstable hemodynamic, ischemic cardiac symptoms/signs, and uncontrolled arrhythmia were instructed to immediately terminate exercise training.

SUMMARY:
BACKGROUND Global burdens of heart failure (HF) are increasing in modern societies. High-intensity interval training (HIIT) increases peak oxygen consumption (VO2peak) in HF patients, which was hypothesized to improve the survival of HF patients.

OBJECTIVES The cohort study aimed to highlight the effect of HIIT on long-term survivals of HF patients.

METHODS 329 HF patients, enrolled between 2009 and 2016, received multidisciplinary disease management program (MDP). They had cardiopulmonary exercise test for peak exercise capacity (VO2peak), echocardiographic examination for left ventricular ejection fraction (LVEF), LV end-diastolic diameter (LVEDD), and LV end-systolic diameter (LVESD), b-type natriuretic peptide (BNP), and quality of life questionnaire. HF patients with LVEF≤ 40% (HFrEF) and HF patients with LVEF> 40% (HFpEF) underwent≥ 36 times of HIIT. HFrEF and HFpEF patients were classified as the MDP group. Generalized estimating equation (GEE) was used to estimate the interaction between time and VO2peak, LVEF, LVEDD, LVESD, and BNP during the follow-up. Survival analysis was conducted to assess effects of HIIT on the long-term survival of HF during at end of the study.

ELIGIBILITY:
Inclusion Criteria:

From January 1st, 2009 to December 31st, 2016, HF patients, defined according to the European society of cardiology, with stable clinical status greater than 4 weeks after optimal treatment were enrolled in the study.

Exclusion Criteria:

Those, who were ≥ 80 years and < 20 years, unable to perform exercise caused by other non-cardiac disease, pregnant, future cardiac transplantation within 6 months, uncompensated HF patients, pacemaker patients, and renal patients with estimated glomerular filtration rate < 30 ml/min/1.73m2, were not candidates in the study. Patients had absolute contraindications for cardiopulmonary exercise test (CPET) and aerobic activities, suggested by the American College of Sports Medicine (ACSM), were also excluded in the study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Baseline information of all eligible candidates, including age, gender, body mass index (BMI), and disease duration were recorded. Serum low-density lipoprotein (LDL), creatinine (Cre), high sensitivity C-reactive protein (hs-CRP), glycohemoglobin (Hba1c), and b-type natriuretic peptide (BNP) were evaluated during the follow-up. Each blood sampling for BNP analysis and short form-36 health survey (SF-36) of physical component score (PCS) and mental component score (MCS) for qualities of life were performed just before each cardiopulmonary exercise test and echocardiographic examination.
Sampling Method: Non-Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
all-cause death | 2009/1/1 to 2016/12/31
  Any mortality during the study period
all-cause re-admission | 2009/1/1 to 2016/12/31
  Any re-admission during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Chin Hsu, MD, PhD, Principal Investigator — Dept. of PM&R, Keelung Chang Gung Memorial Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Fu TC, Wang CH, Lin PS, Hsu CC, Cherng WJ, Huang SC, Liu MH, Chiang CL, Wang JS. Aerobic interval training improves oxygen uptake efficiency by enhancing cerebral and muscular hemodynamics in patients with heart failure. Int J Cardiol. 2013 Jul 15;167(1):41-50. doi: 10.1016/j.ijcard.2011.11.086. Epub 2011 Dec 22. PMID 22197120
- [Result] Lee MF, Chen WS, Fu TC, Liu MH, Wang JS, Hsu CC, Huang YY, Cherng WJ, Wang CH. Non-invasive cardiac index monitoring during cardiopulmonary functional testing provides additional prognostic value in patients after acute heart failure. Int Heart J. 2012;53(6):364-9. doi: 10.1536/ihj.53.364. PMID 23258137